CLINICAL TRIAL: NCT07313033
Title: [68]GA-FAPI-46 PET/CT for the Diagnosis of Metastatic Lesions in Patients With Lobular Breast Cancer (ICL)
Acronym: FAPI-CL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL23_1133; 2025-524897-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Lobular Carcinoma; Breast Cancer
Keywords: lobular carcinoma; medical imaging at [68]GA-FAPI-46 PET scan; oncology; gynecology
MeSH Terms: conditions — Carcinoma, Lobular; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will carry out 2 examinations [18F]-FDG and [68]GA-FAPI-46 PET scan and the gold standard will be histology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental): Adult patients with infiltrating lobular carcinomas. Patients must have had a negative or doubtful 18F-FDG PET/CT scan as part of their routine care pathway
  Interventions: Other: [68]GA-FAPI-46 PET scan

INTERVENTIONS:
Other: [68]GA-FAPI-46 PET scan — Realization of a [68]GA-FAPI-46 PET scan to detect at least one [68]GA-FAPI positive lesion (confirmed by histology)

SUMMARY:
Invasive squamous cell carcinoma (ISCC) represents 5 to 15% of breast cancers. Despite the rarity of this pathology, the number of patients with Invasive squamous cell carcinoma treated at HCL is significant.

Patients at risk of metastasis are usually referred to the HCL Nuclear Medicine departments to perform positron emission tomography - computed tomography (PET/CT) with [18]F-FDG as an extension assessment. The investigators know that [18]F-FDG PET/CT has limited diagnostic performance for assessing the extent of breast cancer with a sensitivity of 66-96% for all histologies combined. For the ISCC, these performances are even lower with average Standard Uptake Value (SUV) values of 3.4 [2.8-3.9] versus 6.6 [4.8-9.7] for the others histological types of breast cancer. False negatives in [18]F-FDG PET/CT are due to an insufficient osteoblastic and immune response in the tumor stroma. Avril & al. showed 65.2% false negatives with [18]F-FDG PET/CT for ISCC. This is why the search for new imaging techniques in this indication is particularly relevant.

Targeting fibroblast activation protein (FAP), a type II membrane glycoprotein belonging to the dipeptidyl peptidase-4 family, is a promising strategy for imaging tumor stroma, particularly in epithelial carcinomas .

The investigators would like to compare the [18]F-FDG PET/CT technique currently used to this new emerging modality.

The investigators hypothesize superior diagnostic performance of [68]Ga-FAPI PET/CT compared to [18]F-FDG PET/CT for the assessment of ISCC extension, with a gold standard histological.

The investigators translate this into the hypothesis of finding 30% of positive FAPI PET when the [18F]FDG PET/CT is negative or doubtful.

The advantage of this project and this new imaging modality is to not undertreat patients wrongly classified as non-metastatic. The investigators therefore wish to offer [68]Ga-FAPI PET/CT to patients with negative [18]F-FDG PET/CT.

The FAPICL project constitutes a seed project before a larger structuring study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old),
* Beneficiary or entitled to a social security system;
* Patient having agreed to participate in the study and signed written informed consent;
* 18F-FDG PET/CT performed as part of the assessment of extension of an infiltrating lobular carcinoma, the result of which is negative or doubtful on at least one lesion.

Exclusion Criteria:

* Pregnant, parturient or breastfeeding women. A pregnancy test before inclusion will be carried out for women of childbearing age.
* Persons deprived of liberty by a judicial or administrative decision
* People receiving psychiatric care
* People admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Subjects participating in another interventional research including an exclusion period still ongoing at inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients for whom at least one secondary lesion is demonstrated in [68]Ga-FAPI and confirmed by histology, when [18]F-FDG PET/CT is negative | 6 weeks

SECONDARY OUTCOMES:
Average number per patient of lesions demonstrated in [68]Ga-FAPI, not seen in [18F]-FDG | 6 weeks
  This criteria will be collected when the imaging is read by a nuclear physician.
Number of lesions positive on histology, among the lesions visualized on PET/CT with [68]Ga-FAPI (and in the case of negative histology, identify the differential diagnoses) | 6 weeks
  This criteria will be collected at the time of publication of the histological report of the suspicious lesion detected.
Evaluate the Positive Predictive Value of [68]Ga-FAPI PET/CT at the patient level, in patients negative on [18]F-FDG PET/CT | 6 weeks
  This criterion will be collected at the time of publication of the histological report of the suspicious lesion detected.
Analyze the semi-quantitative values of the PET signal by describing the [68Ga]-FAPI lesional SUVs, compared to the vascular and hepatic background | 6 weeks
  SUVmax bw lesion, SUVmax liver, SUVmax aorta will be collected at the time of reading the imaging by a nuclear physician, for each suspicious lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Lyon sud Hospital center - Hospices Civils de Lyon, Lyon, France